CLINICAL TRIAL: NCT01460173
Title: Aufmerksamkeitstest Mittels Fahrsimulation Bei Normalpersonen Und Patienten Mit Obstruktivem Schlafapnoesyndrom
Brief Title: Divided Attention Steering Simulator Alertness Test
Acronym: DASS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut für Pneumologie Hagen Ambrock eV (Industry)
Collaborators: Reinhard Löwenstein-Stiftung (Unknown)
Responsible Party: Principal Investigator, Georg Nilius, Head of pneumological department of Helios Klinik Hagen Ambrock, Helios Klinik Ambrock
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: DASS2011
Record Dates: First submitted 2011-10-25; First posted 2011-10-26 (Estimated); Last update posted 2012-09-25 (Estimated); Status verified 2012-09

CONDITIONS: Sleep Apnea, Obstructive
Keywords: alertness test; sleepiness; vigilance; Sleep Apnea, Obstructive
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleepiness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normal subjects (Other)
  Interventions: Other: Divided Attention Steering Simulator (DASS)
- OSA Patients (Other)
  Interventions: Other: Divided Attention Steering Simulator (DASS)

INTERVENTIONS:
Other: Divided Attention Steering Simulator (DASS) — Half-hour divided attention test with steering wheel after 5 to 10 minutes of practice. Completion of three questionnaires (ESS, Young, Berlin Questionnaire).

SUMMARY:
Driving simulator programmes are used under a wide range of conditions, and a correlation of driving performance and real accident risks in patients with obstructive sleep apnoea syndrome(OSAS)could be shown. The most frequently used driving simulator is the Divided Attention Steering Simulator (DASS) of Stowood Scientific Instruments Ltd. (SSI). Until today there are no reference levels with regards to sex and age in existence. To define the boundaries of normality age and sex reference values are to be generated and compared to values of patients with OSAS.

50 male and 50 female healthy subjects (10 of each age decade between 20 and 70 years) will perform the DASS for 30 minutes. In the other arm 100 OSAS Patients will perform the test as well. A better differentiation of pathologic driving performance and response times of OSAS patients should be possible with new reference levels.

DETAILED DESCRIPTION:
The DASS programme records several data, including mean and absloute errors and standard deviations from centre and curve.

Additionally the response time to a randomly appearing target number is recorded (divided attention).

The standard deviation (curve) is the difference between the steering angle and the road angle. Standard deviation (centre) is the standard deviation of the centre of the car from the centre of the road.

Steering performance is quantified as the standard deviation of the error from a theoretical perfect path.

The secondary task of the divided attention test is to respond to a randomly appearing target number at the sides of the monitor while trying to keep the car in the centre of the road.

Average Reaction time is the average time (in seconds) it takes the subject to respond to the target numbers.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects

   * capability of giving consent
   * ESS (Epworth Sleepiness scale) score less than 9
   * Holding a driving license
2. Patients

   * diagnostic OSAS
   * capability of giving consent
   * Holding a driving licence

Exclusion Criteria:

1. Healthy subjects

   * suspected OSAS, any observed sleep disorders or snoring
   * acute cardial, pulmonal oder neurological disease
2. Patients - acute cardial, pulmonal oder neurological disease

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2011-02; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Standard deviations | 30 minutes
  Steering performance is quantified as the standard deviation of the error from a theoretical perfect path.

SECONDARY OUTCOMES:
Reaction time | 30 min
  Reaction time to randomly appearing target numbers to which the subject has to respond.

CONTACTS AND LOCATIONS:
Overall Officials: Georg Nilius, MD, Principal Investigator — Helios Klinik Hagen Ambrock
Locations (1):
- Helios Klinik Hagen Ambrock, Hagen, North Rhine-Westphalia, Germany